CLINICAL TRIAL: NCT04751279
Title: Expression and Role of the JAK/STAT Pathway in Sarcoidosis Granuloma Cells
Acronym: JAK-SARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201205; 2020-A02330-39 (Other: IDRCB)
Record Dates: First submitted 2021-01-29; First posted 2021-02-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sarcoidosis; JAK-STAT Pathway Deregulation
Keywords: Sarcoidosis; JAK/STAT
MeSH Terms: conditions — Sarcoidosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with pulmonary sarcoidosis without signs of chest activity and recent diagnosis (<5 years): Patients with pulmonary sarcoidosis without signs of chest activity (Benamore score <2) and recent diagnosis (<5 years)
  Interventions: Other: Blood sample
- Patients with pulmonary sarcoidosis with signs of chest activity and recent diagnosis (<5 years: Patients with pulmonary sarcoidosis with signs of chest activity (Benamore score ≥2) and recent diagnosis (<5 years)
  Interventions: Other: Blood sample
- Patients with pulmonary sarcoidosis without signs of activity , persistent form (>5 years): Patients with pulmonary sarcoidosis without signs of activity (Benamore score <2), persistent form (>5 years)
  Interventions: Other: Blood sample
- Patients with pulmonary sarcoidosis with signs of chest activity , persistent form (>5 years): Patients with pulmonary sarcoidosis with signs of chest activity (Benamore score ≥2), persistent form (>5 years)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample collection of 5 blood sample at the inclusion in the study the samle consite of 5 tubesEthylene Diamine Tetra Acetate (ADTA) of 7 ml

SUMMARY:
Recent studies suggest that the JAK/STAT signaling pathway constitutes a new step in the clinical and therapeutic progress of sarcoidosis. Further investigations are necessary to identify the most suitable patients to receive treatment targeting this pathway, in particular in cases of severe sarcoidosis refractory to the various therapeutic lines.

DETAILED DESCRIPTION:
The investigators hypothesize that the JAK/STAT signaling pathway constitutes a new step in the clinical and therapeutic progress of sarcoidosis, in particular in cases of severe sarcoidosis refractory to the various therapeutic lines. The main objective of this proposal is to evaluate the presence and stage of activation of the JAK/STAT pathway in PBMCs from inactive and active sarcoidosis patients. The second objective will be to determine the role of the JAK/STAT pathway in the formation and maintenance of granulomas and their association with the severity of sarcoidosis and fibrogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of mediastinopulmonary sarcoidosis made according to ATS / ERS / WASOG criteria
* Or patient suspected of having mediastino-pulmonary sarcoidosis, without any other probable causal factor identified on the usual standard examination at the time of the sample with the need for diagnostic confirmation at the end of the study according to the criteria of the ATS / ERS / WASOG
* Sarcoidosis with stage 1 to 4 pulmonary involvement
* Patients who had a chest CT scan in the 6 months preceding the sample. Examination carried out as part of routine care

Exclusion Criteria:

* Pregnancy.
* Opposition expressed to participation in the study.
* Patients on State Medical Aid.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mediastino-pulmonary sarcoidosis receiving or not receiving treatment for their sarcoidosis. Subjects treated for their sarcoidosis (corticosteroids and/or immunosuppressants) are not excluded because of two recent cases reported of multi-treated patients in which an involvement of the JAK/STAT pathway was demonstrated.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
JAK/STAT familly numbers protein expression in PBMCs | 1 year after inclusion
  Evaluation will be carried out by:
  - studying the expression of members of the JAK/STAT pathway, the expression of cytokines and chemokines phagocytosis and macrophage differentiation the expression of cytokines and chemokines

CONTACTS AND LOCATIONS:
Overall Officials: Florence JENY, MD, Principal Investigator — Assistance Publique - Hôpitaux Paris
Locations (1):
- Service de pneumologie Hôpital Avicenne, Bobigny, France

REFERENCES:
- [Background] Rotenberg C, Besnard V, Brillet PY, Giraudier S, Nunes H, Valeyre D. Dramatic response of refractory sarcoidosis under ruxolitinib in a patient with associated JAK2-mutated polycythemia. Eur Respir J. 2018 Dec 20;52(6):1801482. doi: 10.1183/13993003.01482-2018. Print 2018 Dec. No abstract available. PMID 30361243